CLINICAL TRIAL: NCT06820801
Title: Assessment of Pelvic Floor Muscles Strength and Function After Radiotherapy Treatment in Women With Pelvic Cancers
Brief Title: Assessment of PFM Strength and Function After Radiotherapy Treatment in Women With Pelvic Cancers
Acronym: PFM
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Hassan Khalled Abotaleb, Eman Abotaleb, Cairo University
Other Study IDs: 0237617692
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Muscle Strength and Function
Keywords: pelvic floor muscles - radiotherapy - pelvic cancers
MeSH Terms: interventions — Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: pelvic floor muscles strength and function — using pressure perineometer to evaluate pelvic floor muscles strength and using PFDI to evaluate pelvic floor muscles function

SUMMARY:
Assessment the effect of radiotherapy treatment on pelvic floor muscles in women with pelvic cancers

DETAILED DESCRIPTION:
Evaluate the impact of radiotherapy treament on pelvic floor muscles strength and function in women with cervical and rectal cancers

ELIGIBILITY:
Inclusion Criteria:

* women between 30 -50 years old
* diagnosed with cervix or rectal cancers
* married
* will be treated with preoperative radiotherapy for at least 5 weeks
* had not any pelvic operations in the past

Exclusion Criteria:

* un married women
* Age below 30 or above 50 years old
* has another type of pelvic tumors
* has any metastasis
* had any pelvic surgeries
* will be treated with short course radiotherapy

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: women aged between 30 and 50 years old diagnosed with cervix or rectal cancers and will be treated with preoperative radiotherapy for 5 weeks
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
PFM strength and function | 3 months
  Pelvic floor muscles strength and function

CONTACTS AND LOCATIONS:
Overall Officials: Elham Shahat Hassan, Lecturer of physical therapy, Study Director
Locations (1):
- Elahrar oncology center and zagazeg university oncology center, Zagazeg, Alsharkia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided